CLINICAL TRIAL: NCT05632068
Title: The Efficacy of Xian-Hua-Cha for Improving Hyperlipidemia Among Obese Population: a Crossover Trial
Brief Title: Xian-Hua-Cha for Relieving Hyperlipidemia With Obesity
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: KMRPC5M001
Record Dates: First submitted 2022-11-20; First posted 2022-11-30 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2023-11

CONDITIONS: Hyperlipidemias; Obesity; Body Fat Disorder
Keywords: Chinese herbal medicine; Xian-Hua-Cha; hyperlipidemia; obesity; body fat
MeSH Terms: conditions — Hyperlipidemias; Obesity

STUDY DESIGN:
Intervention Model Description: All eligible subjects will be allocated randomly to 2 groups. Each group will have a 7-month course, including 3-month XHC treatment and 3-month no XHC treatment period (control). One month washout period will be arranged between these two 3-month treatment periods.
Masking Description: A number generated by random sequence before enrollment will be assigned to each subject to separate all subjects to two groups. Diet education/monitoring will be given with or without XHC depending the phase of trial course. Since XHC is a mixture of herbal products and difficult to make proper placebo, we adopt the crossover with open-label design in this study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xian-Hua-Cha (XHC) group (Experimental): Xian-Hua-Cha (XHC) 520 mL, twice a day will be given with diet education/monitoring program for this group for 3 months, followed by one-month wash-out period and a 3-month period with diet education/monitor program alone.
  Interventions: Drug: Xian-Hua-Cha
- Control group (No Intervention): Diet education/monitoring program (500 kcal lower than estimated total energy expenditure of each subject) will be given to each subject for 3 months first, followed by one month wash-out period and a 3-month period of Xian-Hua-Cha (XHC) 520 mL, twice a day, intervention course.

INTERVENTIONS:
Drug: Xian-Hua-Cha — Zizyphus jujuba Mill., Nelumbo nucifera Gaertn, Citrus reticulata Blanco, Rosa rugosa Thunb., Cassia obtusifolia L., Stevioside, resistant starch, and water
  Other Names: XHC
  Arms: Xian-Hua-Cha (XHC) group

SUMMARY:
In the past decades, lipid and body fat disorders become a serious global healthcare issue, especially among the obese population. The aim of this study is to include 100 selected patients with BMI higher than 27 and hyperlipidemia, and a crossover design is used to explore the efficacy of "Xian-Hua-Cha (XHC)" on relieving hyperlipidemia among obese patient. For this purpose, the changes of patients' body weight, body fat and the metabolic parameter including blood sugar, cholesterol, triglyceride are analyzed in the end of this study.

DETAILED DESCRIPTION:
Recently, there are more and more studies show the natural herbal products can improve obesity and related metabolic disorders through changing the body composition and even body weight, but most of the studies are still at the phase of animal studies.

In the ancient Chinese medical book Danxi's mastery of medicine mentioned "Overweight people often have phlegm." From the past observational study, obesity is related phlegm, and the recent concept shows that obesity is a chronic inflammation disease. Therefore, we combined phlegm removal herbal medicine and Chinese medicine for clearing heat and detoxifying together for obese patients with lipid disorders in clinical practice. The aim of this study is to include 100 selected patients with BMI higher than 27 and hyperlipidemia, and a crossover design is used to analyze the efficacy of "Xian-Hua-Cha (XHC)" on relieving hyperlipidemia among the obese population. For this reason, the changes of patients' body weight, body fat and the metabolic parameter including blood sugar, cholesterol, triglyceride are collected for analysis. Besides, we also record adverse effects from taking XHC to assess the safety of XHC.

ELIGIBILITY:
Inclusion Criteria:

1. BMI ≧ 27kg/m2
2. Total cholesterol > 200 mg/dL or LDL > 130 mg/dL or triglyceride > 150 mg/dL
3. Age ≧ 20 years and < 75 years
4. No recognition difficulties
5. Willing to sign inform consent and comply to protocol

Exclusion Criteria:

1. Pregnant or breast-feeding women
2. Endocrine disorders (uncontrolled hypo/hyperthyroidism, adrenal gland disorder)
3. Diagnosis of neurologic or psychiatric diseases
4. Liver or renal dysfunction (AST/ALT higher than 3 times of upper normal limits; eGFR < 60 mL/min/1.73 m2)
5. Acute stress condition (severe infection, receive major surgery in the recent 1 month)
6. Vision, or hearing impairment
7. With other clinical trial medication
8. With medication for obesity or hyperlipidemia in the recent 1 month
9. Heavy smoker, alcoholism or substance abuse
10. Severe organ dysfunction: malignancies, autoimmune diseases

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-12-13 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes on serum lipid profile | 1-2 weeks before trial starting (day 0), 12 (first period), 16 (wash-out), and 28 week (second period)
  The changes on serum triglyceride, total cholesterol, LDL (low-density lipoprotein) cholesterol, and HDL (high-density lipoprotein) cholesterol.

SECONDARY OUTCOMES:
Changes on body weight | 1-2 weeks before trial starting (day 0), 12 (first period), 16 (wash-out), and 28 week (second period)
  The changes on body weight and body mass index (BMI)
Changes on body fat composition | 1-2 weeks before trial starting (day 0), 12 (first period), 16 (wash-out), and 28 week (second period)
  The changes on percentage of body fat and visceral fat, waist to hip ratio, and waistline.

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Linkou and Taoyuan branch, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
Sharing IPD is based on request, and the release of IPD must be approved by the Institutional Review Board of the Chang Gung Medical Foundation

REFERENCES:
- [Background] Hou HI, Chen HY, Lu JJ, Chang SC, Li HY, Jiang KH, Chen JL. The Relationships between Leptin, Genotype, and Chinese Medicine Body Constitution for Obesity. Evid Based Complement Alternat Med. 2021 May 7;2021:5510552. doi: 10.1155/2021/5510552. eCollection 2021. PMID 34055005
- [Background] Liao YN, Chen HY, Yang CW, Lee PW, Hsu CY, Huang YT, Yang TH. Chinese herbal medicine is associated with higher body weight reduction than liraglutide among the obese population: A real-world comparative cohort study. Front Pharmacol. 2022 Sep 9;13:978814. doi: 10.3389/fphar.2022.978814. eCollection 2022. PMID 36160410